CLINICAL TRIAL: NCT03591471
Title: Demonstrated Study on Children Henoch-Schönlein Purpura Nephritis With Multistep Treatment of Traditional Chinese Medicine Combined Disease and Syndrome Differentiation
Brief Title: Study on Children Henoch-Schönlein Purpura Nephritis With TCM Multistep Treatment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: Peking University First Hospital (Other); Children's Hospital of Fudan University (Other); Shanghai Children's Hospital (Other); Chengdu University of Traditional Chinese Medicine (Other); Affiliated Hospital of Yunnan University of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCM for Children HSPN; 2013BAI02B07 (Other Grant/Funding Number: National Science & Technology Support)
Record Dates: First submitted 2014-12-09; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Henoch-Schönlein Purpura Nephritis
Keywords: Children，; Henoch-Schönlein Purpura Nephritis; Integrated and Stepped Treatment in TCM
MeSH Terms: interventions — Prednisone; benazepril; Dipyridamole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM multistep therapy (Experimental): Light HSPN:1.Glycosides Of Tripterygium Wilfordii Hook(GTW): initial dosage is 1.5mg/kg/d(4 weeks),continued with 1mg/kg/d(8 weeks),12weeks in total. Severe HSPN:1.GTW:the initial dosage is 2mg/kg/d(2 weeks), continued with 1.5mg/kg/d(2 weeks) and 1mg/kg/d(8 weeks); 12weeks in total.
  On the above base,Sulfotanshinone Sodium Injection(1mg/kg/d,2weeks) and Qingrezhixue granules(a nosocomial preparation) combined with Chinese herbs(12weeks) based on TCM syndrome differentiation are taken at the same time.
  Interventions: Drug: Glycosides Of Tripterygium Wilfordii Hook(GTW); Drug: Sulfotanshinone Sodium Injection; Drug: Chinese herbs based on syndrome differentiation
- Routine medicine (Active Comparator): Light HSPN:1.Lotensin: 5-10mg/d,12weeks; 2.Low Molecular Weight Heparin(LMWH):100u/kg,2weeks;3.Dipyridamole:3mg/kg/d,Tid,12weeks.4.Chinese medicine placebo,12weeks.
  Severe HSPN:Add pednisone on the treatment of Light HSPN,and gradually reduce the dosage in 12 weeks,the initial dosage is 2mg/kg/d(maximum to 30mg,4 weeks),continue to reduce the dosage until discontinued（Reduce the dosage at the rate of 5mg every other day in 4-8 weeks，then reduce the dosage at the rate of 5-10mg per week in 8-12weeks）
  Interventions: Drug: Prednisone Acetate Tablets; Drug: Benazepril Hydrochloride Tablets; Drug: Low Molecular Weight Heparin Calcium Injection; Drug: Dipyridamole Tab 25 MG; Drug: Chinese medicine placebo

INTERVENTIONS:
Drug: Glycosides Of Tripterygium Wilfordii Hook(GTW) — For severe HSPN GTW is 2mg/kg/d for the first 2 weeks , continued with 1.5mg/kg/d (maximum to 90mg/d) for another 2 weeks; For light HSPN GTW is 1.5mg/kg/d(maximum to 90mg/d) for 4 weeks.
  Both the 2 types are continued with 1mg/kg/d of GTW for another 4 weeks . Besides,Sulfotanshinone Sodium Injection,Qingrezhixue graunles,Chinese herbs by syndrome differentiation are plused at the same time
  Arms: TCM multistep therapy
Drug: Sulfotanshinone Sodium Injection — Intravenous drip of Sulfotanshinone Sodium Injection with the dosage of 1mg/kg/d(maximum to 50mg), combined with 100-250ml 5% Glucose Solution (G.S) for 2 weeks in both the light and serious type of TCM group.
  Arms: TCM multistep therapy
Drug: Chinese herbs based on syndrome differentiation — For both the light and serious type of HSPN in TCM group,five traditional Chinese medicine patterns of syndrome are classified on the main pathogenesis "Blood Stasis": based on Qingre Zhixue granule,for wind-heat complicated with blood stasis, add Forsythia, Honeysuckle,;for blood-heat complicated with blood stasis,add Buffalo horn,Comfrey; for yin deficiency complicated with blood stasis, add Rhizoma anemarrhenae,Cortex phellodendri;for both qi and yin deficiency complicated with blood stasis,add Astragalus, Heterophylla;for damp-heat complicated with blood stasis,add Scutellaria baicalensis,Lalang Grass Rhizome.
  Arms: TCM multistep therapy
Drug: Prednisone Acetate Tablets — Prednisone Acetate Tablets are necessary for serious HSPN in controlled group,the initial dosage is 2mg/kg/d(maximum to 30mg,4 weeks),continue to reduce the dosage until discontinued（Reduce the dosage at the rate of 5mg every other day in 4-8 weeks，then reduce the dosage at the rate of 5-10mg per week in 8-12weeks）
  Arms: Routine medicine
Drug: Benazepril Hydrochloride Tablets — In controlled group, Benazepril Hydrochloride Tablets are used for both the light and serious type with the dosage of 5-10mg/d(10mg/d for children with weight above 30kg) ,12 weeks in total.
  Other Names: Lotensin
  Arms: Routine medicine
Drug: Low Molecular Weight Heparin Calcium Injection — In controlled group,Low Molecular Weight Heparin Calcium Injection are used for both the light and serious type with the dosage of 100u/kg/d by hypodermic injection for 2 weeks
  Arms: Routine medicine
Drug: Dipyridamole Tab 25 MG — In controlled group,Dipyridamole Tab 25 MG are used for both the light and serious type of HSPN with the dosage of 3mg/kg/d ,3 times a day,12 weeks in total.
  Other Names: Persantine
  Arms: Routine medicine
Drug: Chinese medicine placebo — In controlled group,take a potential necessary for patients who come to the hospital of TCM to take traditional Chinese medicine in consideration, we add the traditional Chinese medicine placebo in controlled group.
  Arms: Routine medicine

SUMMARY:
The purpose of this study is to determine the optimum dosage and application method of Glycosides Of Tripterygium Wilfordii Hook(GTW) for Henoch-Schönlein Purpura Nephritis(HSPN) in children, and develop into the normal treatment protocols for Henoch-Schönlein Purpura Nephritis in children.

DETAILED DESCRIPTION:
Based on Chinese Eleventh Five-year Plan for Science and Technology Program, this study follows a large-sample multicenter centerrandom open-label controlled perspective method, enrolls HSPN children with hematuria associated with proteinuria and isolated proteinuria from 2 to 18 years of age, classifys five traditional Chinese medicine patterns of syndrome: wind-heat complicated with blood stasis, blood-heat complicated with blood stasis, yin deficiency complicated with blood stasis, both qi and yin deficiency complicated with blood stasis,damp-heat complicated with blood stasis. For TCM group,according to the severity of HSPN, stepped treatment should be taken. The initial dosage of GTW for severe HSPN is 2mg/kg/d, continued with 1.5mg/kg/d and 1mg/kg/d; The initial dosage of GTW for light HSPN is 1.5mg/kg/d, continued with 1mg/kg/d. On the above base, the comprehensive treatment are taken combined with TCM syndrome differentiation, medicated with Sulfotanshinone Sodium Injection.For controlled group,the treatment for severe HSPN is prednisone combined with heparin plus lotensin and dipyridamole tablets;for light HSPN is heparin plus lotensin and dipyridamole tablets.12 weeks after treatment, the third-party statistics evaluate the efficacy and effect,and a follow-up lasting 36 weeks will go on.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Henoch-Schönlein Purpura Nephritis Disease
* Age form 2-18 years old
* Disease onset within 2 months

Exclusion Criteria:

* Nephritis not causing by HSPN
* Being alergic to the medicine in the treatment
* No compliance

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
24-hour urinary protein quantity | Changes in the quantity of urinary protein at week 1、week2、week 4、week6、week8、week10 and week12 of the treatment phase and at week16、week20、week24、week28、week32、week36、week40、week44、week48 of the follow-up phase compared with baseline
  24-hour urinary protein is the most important and direct indicators of therapeutic effect,so this clinical lab index should be reccord at every point during treatment and follow-up,17 times in total.

SECONDARY OUTCOMES:
Urine red blood cells | Changes in the quantity of urinary protein at week 1、week2、week 4、week6、week8、week10 and week12 of the treatment phase and at week16、week20、week24、week28、week32、week36、week40、week44、week48 of the follow-up phase compared with baseline
  Compared to 24-hour urinary protein,urine red blood cells count is a secondary indicator to reflect therapeutic effect because urine red blood cells recede more slowly than protein,this clinical lab index should also be reccorded at every point during treatment and follow-up,17 times in total.

OTHER OUTCOMES:
The white blood cell count(WBC) in the blood | Week0(before treatment),week1、week2、week4、week6、week8、week10 and week12 of the treatment phase and week16、week20、week24、week28、week32、week36、week40、week44、week48 of the follow-up phase
  There is a potential risk of abnormality in the blood system in terms of leukocyte counts after taking immunosuppressor or prednison. Leukocyte count should be recorded in total of 17 times during and after treatment through routine blood tests.
The platelet count(PLT) in the blood | Week0(before treatment),week1、week2、week4、week6、week8、week10 and week12 of the treatment phase and week16、week20、week24、week28、week32、week36、week40、week44、week48 of the follow-up phase
  There is a potential risk of abnormality in the blood system in terms of platelet counts after taking immunosuppressor or prednison. Platelet count should be recorded in total of 17 times during and after treatment through routine blood tests.
Glutamate alanine transferase(ALT) in the blood | Week0(before treatment)，week1、week2、week4、week8、week12 of the treatment phase and week20、week28、week36、week44、week48 of the follow-up phase
  There is a potential risk of dysfunction in liver after using any drug. As one of the indicators of liver damage,the test of ALT should be taken in total of 11 times during and after treatment through a liver function test by taking blood from vein.
Glutamate aspartate transferase(AST) in the blood | Week0(before treatment)，week1、week2、week4、week8、week12 of the treatment phase and week20、week28、week36、week44、week48 of the follow-up phase
  There is a potential risk of dysfunction in liver after using any drug. As one of the indicators of liver damage,the test of AST should be taken in total of 11 times during and after treatment through a liver function test by taking blood from vein.
Serum Creatinine(Scr) | Week0(before treatment)，week1、week2、week4、week8、week12 of the treatment phase and week20、week28、week36、week44、week48 of the follow-up phase
  There is a potential risk of dysfunction in kidney after using any drug. As an indicator of kidney damage,the test of Cr should be taken in total of 11 times during and after treatment through a kidney function test by taking blood from vein.
Blood Urea Nitrogen(BUN) | Week0(before treatment)，week1、week2、week4、week8、week12 of the treatment phase and week20、week28、week36、week44、week48 of the follow-up phase
  There is a potential risk of dysfunction in kidney after using any drug. As an indicator of kidney damage，the test of BUN should be taken in total of 11 times during and after treatment through a kidney function test by taking blood from vein.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Ding, professor, Principal Investigator — Henan University of Traditonal Chinese Medicine
Locations (2):
- China (2):
  - Children's Hospital, The First Affiliated Hospital of HUTCM, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: Yes
We allow all the data to be made public once the trial finished
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Our data will become availiable from January,2019 and for 10 years

REFERENCES:
- [Derived] Ding Y, Zhang X, Ren X, Zhai W, He L, Liu J, Yao C, Han S, Wang L. Traditional Chinese medicine versus regular therapy in Henoch-Schonlein purpura nephritis in children: study protocol for a randomized controlled trial. Trials. 2019 Aug 29;20(1):538. doi: 10.1186/s13063-019-3484-3. PMID 31464626